CLINICAL TRIAL: NCT05740787
Title: Inflammatory and Neural Correlates of Chemotherapy-Induced Cognitive Impairment: A Pilot Study
Brief Title: Chemotherapy Induced Cognitive Impairment
Acronym: CONCERT
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-028-22
Record Dates: First submitted 2023-02-07; First posted 2023-02-23 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observation only

SUMMARY:
Chemotherapy is toxic and challenges everyone differently. Most chemotherapy side-effects are known and well documented. However, the phenomenon of "chemo fog" also known as "chemobrain" has not been fully investigated and is often based on comments of breast cancer patients attending outpatient clinics during and after their chemotherapy. Changes in thinking ability like lack of concentration, loss of memory and the inability to hold a thought or even a conversation has a significant impact on the lives of breast cancer patients. Without understanding what "chemobrain" is, and what causes it, there is little that doctors can do to help at the moment.

The team proposing this study believe that chemotherapy causes chemicals associated with inflammation to attack parts of the brain that are important for concentration and making new memories. Unfortunately, it is not possible to measure these chemicals directly in the brain, but we believe that a brain scan sensitive to excess iron, a marker of brain inflammation, can help. This project will measure thinking ability, such as memory and concentration, take a blood sample and do a brain scan before, during and after a patient has chemotherapy. We will then look for changes in iron in the brain areas that are important for concentration and memory and compare those to changes in thinking ability and to levels of inflammation chemicals in the blood. This information will be essential to help plan our next step which is to test ways to reduce the effects of "chemobrain".

DETAILED DESCRIPTION:
Ten critical research gaps and translational priorities in breast cancer were identified and published in 2013. One of them (#9) highlighted the need of developing interventions and support to improve the survivorship experience. It is well known that cancer treatment can cause significant long-term effects on a patient's life. Cognitive dysfunction has been recognised as one of those negative effects. The majority of breast cancer patients are living significantly beyond their breast cancer diagnosis. Most of the patients receiving chemotherapy are deemed to be at performance status '0'; fully participating in society, fully active with no restrictions on any activities prior to their cancer diagnosis. These patients are treated with curative intent. It is anticipated for them to fully integrate and return to their everyday life after their breast cancer treatment has been completed. However, for some this is not the case.

Many side effects of chemotherapy, such as fatigue or immune suppression, are well-known but it is less recognised that chemotherapy can cause long-term changes in concentration, memory and learning. This has been referred to as "chemofog". Recent studies suggest that about 15-45% of patients complain about memory and attention problems, lack of concentration, and deficits in multitasking or decision-making following chemotherapy. A number of possible explanations have been proposed for these changes, one is that many chemotherapy drugs are designed to stop cell division. An important part of normal brain function is neurogenesis, the process of creating new neurons, the building blocks of the brain. If cell division is stopped these building blocks can no longer be produced. The hippocampus and striatum are areas critically important to many brain functions. If new neurons are not made, the hippocampus shrinks which is a marker of the memory problems associated with dementia. As well as reducing neurogenesis, chemotherapeutic drugs can also change the balance of important chemicals in the brain called neurotransmitters. This can lead to decreased focus, arousal, and thinking speed. Finally, chemotherapeutic drugs can induce inflammation which can maintain these deficits for years after treatments cease.

Fifty patients will be recruited who have been diagnosed with breast cancer and are having either neoadjuvant or adjuvant chemotherapy as part of their treatment. They will attend the University of Aberdeen research MRI facility on 3 occasions: 1) within 2 weeks of diagnosis, 2) 4 weeks after the last cycle of chemotherapy, 3) 6 months following the end of chemotherapy. Patients on the most common treatment, anthracyclines with or without taxane, will be the focus of this study. A baseline scan before chemotherapy means each patient will be their own control.

During each visit the following will take place:

Brain magnetic resonance imaging: Brain MRI will be performed using a Philips Ingenia dStream 3T scanner and a 32-channel phase-array head coil. The protocol will include structural images (3D T1-weighted, 3D T2-weighted, 3D susceptibility weighted imaging (SWI), fluid attenuated inversion recovery (FLAIR), resting state fMRI (rs-fMRI) and diffusion tensor imaging (DTI). These sequences will allow us measure regional brain volumes and brain functional connectivity and also to see clinically significant features.

Cognitive and general health assessments: 5 individual components of general intelligence, cognitive fatigue, a potential confounder in cognitive testing, depression and anxiety and general health:

1. Digit Symbol Coding to measure information processing speed
2. Mill Hill Vocabulary test used as a measure of acquired verbal intelligence and an estimate of peak cognitive ability
3. Controlled Oral Word Association task used as a measure of verbal fluency
4. The Logical Memory test used to assess

   1. immediate declarative recall
   2. delayed declarative recall (30 min. apart)
5. Matrix Reasoning test, assessing perceptual organisation and visuospatial logic
6. Chalder Fatigue Scale
7. Hospital Anxiety and Depression Scale
8. General Health Questionnaire Blood sample collection: Blood samples will be collected at the time of imaging and cognitive testing to allow high sensitivity ELISA (Enzyme-Linked Immunosorbent Assay) tests for plasma levels of inflammation markers: Total body iron index (sTfR and Ferritin), IL-6, TNF-alpha, IL-1beta, Glutathione Peroxidase-3 (GPX3) activity, Colony-stimulating factor 1 (CSF-1), high-sensitivity c-reactive protein (hsCRP) and F2-isoprostane, a systemic marker of oxidative stress that reflects lipid peroxidation levels. A full blood count will be performed to screen for clinically significant levels of anaemia and immune cell counts.

ELIGIBILITY:
Inclusion Criteria:

* Women and men >18 years
* Diagnosed with HER2 negative breast cancer
* Receiving EC-Taxane or Taxane only based chemotherapy
* Able to communicate in English
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Any patient whose physical condition will preclude them from lying still for the duration of the brain scan.
* pre-excisting mental condition/disability
* Contraindication to magnetic resonance scanning such as an implantable cardiac device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Breast Cancer who have been prescribed adjuvant or neo-adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance late post chemotherapy | 6 months
  General intelligence will be determined with PCA from 5 separate tests to give 'g' general intelligence.
  'g' is scaled to have a mean of 100 and a standard deviation of 15 giving an IQ-like measure of general intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No